CLINICAL TRIAL: NCT05044065
Title: Blood Flow Restriction Exercise in the Perioperative Setting to Prevent the Loss of Muscle Mass in Patients With Pancreatic, Biliary Tract, and Liver Cancer - the PREV-Ex Randomized Controlled Trial
Brief Title: Blood Flow Restriction Exercise in Patients With Pancreatic, Biliary Tract, and Liver Cancer (PREV-Ex)
Acronym: PREV-Ex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other); Norwegian School of Sport Sciences (Other); Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Sara Mijwel, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PREV-Ex
Record Dates: First submitted 2021-08-16; First posted 2021-09-14 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Pancreatic Cancer; Biliary Tract Cancer; Liver Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Biliary Tract Neoplasms; Liver Neoplasms | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise group (Experimental): The experimental group will in addition to standard care receive supervised and home-based exercise training program with a specific focus to induce metabolic stress (blood flow restriction exercise), and protein supplementation to ensure adequate protein intake.
  Interventions: Other: Physical exercise
- Usual care (No Intervention): The control group will in addition to standard care receive protein supplementation to ensure adequate protein intake.

INTERVENTIONS:
Other: Physical exercise — The intervention group will receive an exercise program consisting of a combination of supervised and home-based exercise with a focus to induce metabolic stress (blood flow restriction exercise) during both a pre- and postoperative period consisting of a total of 6-10 weeks. Protein supplementation will be given to exclude insufficient intake.
  Arms: Exercise group

SUMMARY:
In patients with cancer, resistance training appears to be a safe and effective exercise modality to increase both lean muscle mass and strength, as well as attenuates cancer-related fatigue. It may serve as a feasible intervention in these patients to mitigate cachexia, especially if implemented before the onset of cancer cachexia or in a pre-cachectic state. This study is a multicenter randomized controlled trial that will compare a blood flow restricted resistance training intervention during the pre- (prehabilitation) and post-operative (rehabilitation) phase in patients with pancreatic, biliary tract and liver cancer, versus usual care on skeletal muscle and other health-related outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of resectable pancreatic cancer
* Diagnosis of resectable biliary tract cancer (includes cholangiocarcinoma and ampullary cancer)
* Diagnosis of resectable liver cancer
* ECOG (Eastern Cooperative Oncology Group scale) performance status ≤ 2

Exclusion Criteria:

* Serious active infection
* Uncontrolled severe pain
* Severe neurologic or cardiac impairment according ACSM criteria
* Uncontrolled severe respiratory insufficiency as determined by the treating clinician
* Any other contraindications for exercise as determined by the treating physician
* Poor Swedish comprehension
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Skeletal muscle thickness | Change from baseline (T0) to: 1-4 weeks (T1), 4-7 weeks (T2), 10-13 weeks (T3).
  Skeletal muscle thickness (mm) measured through ultrasound
Skeletal muscle cross sectional area | Change from baseline (T0) to: 1-4 weeks (T1), 4-7 weeks (T2), 10-13 weeks (T3).
  Skeletal muscle cross sectional area (um2) measured through ultrasound

SECONDARY OUTCOMES:
Skeletal muscle morphology | Change from baseline (T0) to: 10-13 weeks (T3).
  Skeletal muscle morphology (au) measured through microscopy methods in skeletal muscle biopsies
Skeletal muscle protein levels | Change from baseline (T0) to: 10-13 weeks (T3).
  Skeletal muscle protein levels (au) measured through western blot in skeletal muscle biopsies
Skeletal muscle metabolism | Change from baseline (T0) to: 10-13 weeks (T3).
  Skeletal muscle metabolism (au) measured through biochemical methods in skeletal muscle biopsies
Body lean mass | Change from baseline (T0) to: 1-4 weeks (T1), 4-7 weeks (T2), 10-13 weeks (T3).
  Lean mass (kg) measured through bioimpedance and CT scan
Body fat mass | Change from baseline (T0) to: 1-4 weeks (T1), 4-7 weeks (T2), 10-13 weeks (T3).
  Fat mass (kg) measured through bioimpedance and CT scan
Handgrip strength | Change from baseline (T0) to: 1-4 weeks (T1), 4-7 weeks (T2), 10-13 weeks (T3).
  Maximal handgrip strength (kg) measured through hand dynamometry
Lower limb muscle strength | Change from baseline (T0) to: 1-4 weeks (T1), 4-7 weeks (T2), 10-13 weeks (T3).
  Maximal leg strength (kg) measured through isometric force measurements
Health-related quality of life | Change from baseline (T0) to: 1-4 weeks (T1), 4-7 weeks (T2), 10-13 weeks (T3), 5-6 months (T4).
  Disease specific helath related quality of life measured with The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-C30 (EORTC-QLQ-C30) Summary Score (0-100 points with a higher score indicating a better quality of life)
Physical performance | Change from baseline (T0) to: 1-4 weeks (T1), 4-7 weeks (T2), 10-13 weeks (T3).
  Short Physical Performance Battery (SPPB score points ranging from 0-12 with a higher score indicating a better physical function) measured through handgrip strength test, leg strength test, endurance test
Cancer-related fatigue | Change from baseline (T0) to: 1-4 weeks (T1), 4-7 weeks (T2), 10-13 weeks (T3), 5-6 months (T4).
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Fatigue12 (EORTC-QLQ-FA12) Summary Score (0-100 points with a higher score indicating a better quality of life)
Nutritional status | Change from baseline (T0) to: 1-4 weeks (T1), 4-7 weeks (T2), 10-13 weeks (T3), 5-6 months (T4).
  Subjective Global Assessment Form scores (score ranging between 7 (normal) and 35 (severely malnourished)
Participants' experience of the exercise program | 3 months
  Focus group and individual interviews
Treatment related complications | 4-7 weeks (T2)
  days to recover after surgery will be assessed retrospectively through the patients' medical records.
Hospitalization | 5-6 months (T4)
  days of being hospitalized will be assessed retrospectively through the patients' medical records.
Physical activity | Change from baseline (T0) to: 1-4 weeks (T1), 4-7 weeks (T2), 10-13 weeks (T3), 5-6 months (T4).
  Measured through an activity tracker (hours)
Inflammatory markers | Change from baseline (T0) to: 10-13 weeks (T3)
  Inflammation (au) will be assessed from blood serum and plasma.
Prognostic markers | Change from baseline (T0) to: 10-13 weeks (T3)
  Prognostic markers (au) will be assessed from blood serum and plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Mijwel, PhD, Principal Investigator — Karolinska Institutet
Locations (2):
- Oslo University Hospital, Oslo, Norway
- Karolinska University Hopsital, Stockholm, Sweden

REFERENCES:
- [Derived] Ernst M, Wagner C, Oeser A, Messer S, Wender A, Cryns N, Brockelmann PJ, Holtkamp U, Baumann FT, Wiskemann J, Monsef I, Scherer RW, Mishra SI, Skoetz N. Resistance training for fatigue in people with cancer. Cochrane Database Syst Rev. 2024 Nov 28;11(11):CD015518. doi: 10.1002/14651858.CD015518. PMID 39606939
- [Derived] Anandavadivelan P, Cardinale D, Blomhoff R, Sunde B, Lassen K, Kleive D, Sturesson C, Gilg S, Raastad T, Mijwel S. Blood flow restriction Exercise in the perioperative setting to Prevent loss of muscle mass in patients with pancreatic, biliary tract, and liver cancer: study protocol for the PREV-Ex randomized controlled trial. Trials. 2024 Jun 4;25(1):356. doi: 10.1186/s13063-024-08207-5. PMID 38835083